CLINICAL TRIAL: NCT03255915
Title: Randomized Order, Controlled, Double Blind, Crossover Early Phase 1 Pilot Study to Assess Safety and Pharmacokinetics of a Tenofovir Disoproxil Fumarate and Emtricitabine (TDF-FTC) Releasing IVR Over 28 Days Compared to Placebo
Brief Title: PrEP-Pod-IVR (TDF-FTC/Placebo IVR 28 Day Crossover Study)
Acronym: PrEP-Pod-IVR
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oak Crest Institute of Science (Other)
Collaborators: The Miriam Hospital (Other); Johns Hopkins University (Other); University of California, Los Angeles (Other); University of California, San Diego (Other); Vanderbilt University (Other); The University of Texas Medical Branch, Galveston (Other); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-0131; 1U19AI113048-01 (NIH)
Record Dates: First submitted 2017-07-26; First posted 2017-08-21 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: HIV Prevention
Keywords: HIV Prevention; Intravaginal Ring; Tenofovir Disoproxil Fumarate; Emtricitabine
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: Randomized order, placebo-controlled, double blind, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 will receive the Tenofovir Disoproxil Fumarate (TDF)-Emtricitabine (FTC) pod-IVR for Stage 2 followed by the placebo pod-IVR during Stage 3.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF)-Emtricitabine (FTC); Other: Placebo
- Arm 2 (Experimental): Arm 2 will receive the placebo pod-IVR for Stage 2 followed by the Tenofovir Disoproxil Fumarate (TDF)-Emtricitabine (FTC) pod-IVR during Stage 3.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF)-Emtricitabine (FTC); Other: Placebo

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate (TDF)-Emtricitabine (FTC) — TDF-FTC pod-IVR designed to deliver TDF at a target rate of 1 mg d-1 and FTC at a target rate of 2 mg d-1.
Other: Placebo — A placebo pod-IVR containing microcrystalline cellulose pods.

SUMMARY:
Participants will have a 28-day pre-ring baseline assessment period (Stage 1) followed by randomization to order with 5 participants per study arm. All participants will sequentially receive both study products for 28-days with at least a 2-week washout period between products. Arm 1 will receive the TDF-FTC pod-IVR for Stage 2 followed by the placebo pod-IVR during Stage 3. Arm 2 will receive the placebo pod-IVR for Stage 2 followed by the TDF-FTC pod-IVR during Stage 3. During Stages 2 & 3 participants will also complete brief phone surveys (<3 min), computer-assisted self-interviews (CASIs), and in-depth interviews (IDIs) regarding perceptibility and acceptability. If willing, participants' male sexual partners will be invited to complete IDIs as well.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 through 45 years at screening, verified per site SOP
2. Female participants, born female
3. Not pregnant or breastfeeding
4. Availability to return for all study visits, barring unforeseen circumstances
5. Willing and able to

   * communicate in English
   * provide written informed consent to take part in the study
   * provide adequate locator information, as defined in site SOP
   * complete all required study procedures, including phone surveys, daily vaginal swabs, and reliably store swabs in freezer
6. Must agree

   * not to participate in other concurrent interventional and/or drug trials
   * to use study-provided condoms for vaginal or anal intercourse for the duration of the study
   * to abstain from use of any vaginal products (e.g., lubricants, feminine hygiene products, vaginally administered contraceptive products, sex toys) other than study products for the duration of the study beginning at enrollment Note: Tampons may be used during menses, but must be discontinued 72 hours prior to study visits and for 7 days after biopsy procedures. Menstrual pads will be provided to participants.
   * to abstain from receptive oral, vaginal, or anal intercourse during the first week after each pod-IVR insertion and for 2 days before and 7 days after biopsy procedures
   * to abstain from insertion of anything in the vagina (e.g., tampon, finger, sex toy, lubricants, medication, douche) during the first week after each pod-IVR insertion and for 2 days before and 7 days after biopsy procedures
7. Understands and agrees to local STI reporting requirements
8. HIV-1 seronegative at screening
9. Must be in general good health in the opinion of the investigator
10. Regular menstrual cycles of approximately 21 to 35 days apart with no untreated intermenstrual menstrual bleeding Note: This criterion is not applicable to participants using continuous combination oral contraceptive pills or progestin-only methods (such as Depo-Provera or levonorgestrel-releasing IUD), as the absence of regular menstrual cycles is an expected, normal consequence in this context.
11. Satisfactory cervical Pap result in the 36 calendar months prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies [Addendum 1, Dated November 2007], or if Grade 1 or higher Pap result has had a satisfactory evaluation with no treatment required per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines in the 12 calendar months prior to Enrollment
12. Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation. Acceptable methods include:

    * hormonal methods (except contraceptive vaginal rings)
    * IUD
    * sterilization of participant or partner

    In addition to the criteria listed above, participants who agree to have rectal biopsies collected must meet the following criteria:
13. Must agree to abstain from insertion of anything in the rectum (e.g., finger, sex toy, lubricants, medication, enema) during the first week after each pod-IVR insertion and for 2 days before and 7 days after biopsy procedures

Male sexual partner(s) who meet the following criteria are eligible for inclusion in the study:

1. Age of 18 years or over
2. Has a female sexual partner enrolled in the study
3. Willing and able to

   * communicate in English
   * provide written informed consent to take part in the study
   * provide adequate locator information, as defined in site SOP
   * complete in-depth interview via video conference

Exclusion Criteria:

Individuals who meet any of the following criteria will be excluded from the study:

1. Undergoing or completed gender reassignment
2. Participant reports any of the following at Screening:

   1. Has plans to relocate away from the study site area during the period of study participation
   2. Pregnant, less than 3 months post-partum, or lactating
   3. Intends to become pregnant during the period of study participation
   4. Current or planned use of an IVR
   5. Known HIV-infected partners
   6. Non-therapeutic injection drug use in the 6 months prior to screening
   7. History of autoimmune disease
   8. History of toxic shock syndrome
   9. History of adverse reaction to TDF, FTC, silicone, or microcrystalline cellulose
   10. PrEP or Post-exposure prophylaxis for HIV exposure within 6 months prior to screening
   11. Use of systemic immunomodulatory medications within the 4 weeks prior to the Enrollment
   12. Use of vaginally or rectally administered medications or products (including condoms) containing Nonoxynol-9 (N-9) within the 4 weeks prior to the Enrollment
   13. Participating in another research study involving drugs or medical devices within the 4 weeks or 5 half-lives (if known) prior to the Enrollment
   14. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) within 60 days prior to Enrollment

   Note: Colposcopy and cervical biopsies for evaluation of an abnormal Pap smear as well as IUD removal are not exclusionary
3. Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation:

   1. Heparin, including Lovenox® (enoxaparin sodium)
   2. Warfarin
   3. Plavix® (clopidogrel bisulfate)
   4. Any other drugs that are associated with increased likelihood of bleeding following mucosal biopsy (e.g., daily high dose aspirin, Pradaxa®)
   5. NSAID use for 5 half-lives prior to biopsy (e.g. ibuprofen for 1 day, naproxen for 4 days).
   6. Rectally or vaginally administered medications (including over-the-counter products)
4. History of significant gastrointestinal bleeding in the opinion of the investigator
5. Abnormalities of the cervical, vaginal, or colorectal mucosa, or significant symptom(s), which in the opinion of the clinician represents a contraindication to protocol-required biopsies (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids). Erythema is not exclusionary.

   • Includes any clinically apparent Grade 2 or higher pelvic examination finding (observed by study staff) at Screening or Enrollment, as per the Female Genital Grading Table for Use in Microbicide Studies [Addendum 1, Dated November 2007]
6. At screening: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic bacterial vaginosis, symptomatic vaginal candidiasis, trichomoniasis, chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, pelvic inflammatory disease, genital sores or ulcers, cervicitis, or symptomatic genital warts requiring treatment (i.e., those that cause undue burden or discomfort to the participant).

   Note:
   * An HSV-1 or HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required
   * One re-screening after documented treatment will be allowed
7. Has any of the following laboratory abnormalities at Screening:

   Note: Grade is per Version 2.1 of the DAIDS Toxicity Table
   1. Hemoglobin Grade 1 or higher
   2. Platelet count Grade 1 or higher
   3. International Normalized Ratio (INR) Grade 2 or higher
   4. White blood cell count Grade 2 or higher
   5. Calculated creatinine clearance ≤ 80 mL/minute using the Cockcroft-Gault equation
   6. Grade 2 or higher ALT and/or AST (i.e., ≥ 2.5x the site laboratory upper limit of normal [ULN])
   7. Positive for Hepatitis B surface antigen (HBsAg)
   8. Positive for Hepatitis C antibody (HCV Ab)
8. Has any other condition that, in the opinion of the Principal Investigator or designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Male sexual partner(s) who meet the following criteria are not eligible for inclusion in the study:

1) Female partner did not utilize study product

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Vaginal IVRs releasing TDF-FTC by reports of Adverse Events | From date of enrollment until the date of study completion or date of study withdrawal from any cause, whichever came first, assessed up to 6 months
  Adverse events Grade 2 or higher as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017, Addendum 1 Female Genital Grading Tables for Use in Microbicide Studies (November 2007), and/or Addendum 3 Rectal Grading Table for Use in Microbicide Studies (Clarification dated May 2012) to this table
Characterization of pharmacokinetics of TDF-FTC released by an IVR - plasma | From date of enrollment until the date of study completion or date of study withdrawal from any cause, whichever came first, assessed up to 6 months
  To characterize the local and systemic pharmacokinetics (PK) of TDF-FTC delivered via a pod-IVR, including drug concentration in plasma.
Characterization of pharmacokinetics of TDF-FTC released by an IVR - vagina | From date of enrollment until the date of study completion or date of study withdrawal from any cause, whichever came first, assessed up to 6 months
  To characterize the local and systemic pharmacokinetics (PK) of TDF-FTC delivered via a pod-IVR, including drug concentration in vaginal secretions and tissue.
Characterization of pharmacokinetics of TDF-FTC released by an IVR - rectum | From date of enrollment until the date of study completion or date of study withdrawal from any cause, whichever came first, assessed up to 6 months
  To characterize the local and systemic pharmacokinetics (PK) of TDF-FTC delivered via a pod-IVR, including drug concentration in rectal secretions.

SECONDARY OUTCOMES:
Acceptability of IVR assessed via computer assisted self interviews | 28 days after use of each IVR
  Self-reported attitudes of participants about experience and product attributes via computer assisted self interviews
Acceptability of IVR assessed via in depth interviews | 28 days after use of each IVR
  Self-reported attitudes of participants about experience and product attributes via in depth interviews
Adherence | From date of IVR insertion until the date of IVR removal or date of study withdrawal from any cause, whichever came first, assessed up to 6 months
  Measured by vaginal fluid PK drug levels, vaginal tissue PK drug and drug metabolite levels, and residual drug levels in returned, used pod-IVRs.
Acceptability of IVR assessed via in depth interviews - male partners | 28 days after subject use of each IVR
  Self-reported attitudes of participant's male sexual partner(s) about experience and product attributes via in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Vincent, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Informed Consent Form: Screening Consent (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03255915/ICF_003.pdf
  • Informed Consent Form: Enrollment Consent (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03255915/ICF_004.pdf
  • Informed Consent Form: Male Partner Consent (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03255915/ICF_005.pdf